CLINICAL TRIAL: NCT04257331
Title: Evaluation of a Parent Training Programme for Families of Children With Autism Spectrum Disorder in China: A Mixed-Methods Quasi-Experimental Study
Brief Title: Parent Training to Reduce Behavioral Problems in Children With Autism Spectrum Disorder in China
Acronym: SREIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Beijing Normal University (Other); Beijing Stars and Rain Education Institute for Autism (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R67619/RE001
Record Dates: First submitted 2020-01-30; First posted 2020-02-06 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-04

CONDITIONS: Child Behavior Problem; Autism Spectrum Disorder; Parent-Child Relations; Parenting; Mental Health Issue; Child Abuse; Family Relations
Keywords: Parenting Education; Quasi Experimental Design; Propensity Score Weight
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Stars, Celestial

STUDY DESIGN:
Intervention Model Description: A pragmatic quasi-experimental study will be conducted to examine the effectiveness of the SREIA programme. The study will be conducted within the context of routine services and will involve two consecutive deliveries of the SREIA programme. One hundred families of children with ASD age three to six will be recruited and allocated to the two waves of delivery based on their availability and preference, with 50 families in each wave. Each wave will comprise two versions of the programme that are delivered concurrently, with 30 families in version A and 20 in version B. Participants will be self-selected into either version. The 50 families who choose to participate in the first wave will be the treatment group, and the 50 families in the second wave will service as the waitlist control group.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of parent training and the use of a waitlist control group, it will not be possible to blind participants or facilitators. However, research staff who collect the data will be blinded for the baseline and post-intervention assessment. Data collectors will not be involved in the delivery process and will be trained on the topic of risk of bias. Parents will also be asked not to reveal their allocation condition to outcome data collectors. Process evaluation data will be collected by a separate group of research staff. Given that all families will ultimately receive the training, blinding will not be possible at the follow-up time-points. Blinding will be protected and monitored, while the violation of blinding will be detected and incorporated into the interpretation of results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SREIA group (Experimental): Participants in this arm will be families who attend the first wave of the two rounds of delivery. They will be the intervention group.
  Interventions: Behavioral: Stars and Rain Education Institute for Autism (SREIA) Parent Training Programme
- Waitlist Control (No Intervention): Participants in this arm will be families who attend the second wave of the two rounds of delivery. They will be the control group.

INTERVENTIONS:
Behavioral: Stars and Rain Education Institute for Autism (SREIA) Parent Training Programme — The SREIA program is grounded in applied behavior analysis and developmental theories. It aims to reduce child behavioral problems and promote child development by improving parental attitudes and parenting styles. The program targets parent-child dyads from families of children with ASD aged between three and six years. It is delivered five days a week for 11 weeks. Fourteen two-hour lectures on weekly themes (such as knowledge of ASD, parent-child interaction, and behavior management techniques) are offered throughout the 11 weeks and attended by all participating parents. For the remaining time, additional training in ABA principles and practice are tailored for the different functioning groups. The program offers a combination of individual counselling and group sessions, as well as a mixture of didactic and interactive delivery modes. All sessions are delivered in person. Some sessions are only for parents and others are participated in by both parent and child.
  Arms: SREIA group

SUMMARY:
Objectives The primary objective of this study is to evaluate the effectiveness of the SREIA parent training program for families of children with ASD aged three to six years in mainland China. The study will be conducted within the context of routine service provision and assess the effectiveness of SREIA in reducing child behavioral problems as measured by the Externalizing scale of the Child Behavior Checklist (CBCL) for Ages 1.5-5, in comparison to a waitlist control group.

Secondary objectives include examining the effectiveness of the SREIA program in reducing ASD symptoms and improving parental and familial outcomes including parental knowledge of ASD and ABA techniques, parenting styles, parental mental health (including stress, anxiety and depression), and family functioning.

A process evaluation will be conducted alongside the quasi-experimental trial, the objectives of which are to 1) describe the implementation aspects of the programs with regard to participant involvement, program acceptability, delivery, and sustainability; 2) explore predictors of participant involvement; and 3) examine potential relations between implementation aspects and treatment effects.

Background ASD is associated with elevated levels of child emotional and behavior disturbance, which impair child daily functioning and impose challenges to parenting. The SREIA programme is a group-based parent training in China, that has been delivered since 1993 and reached over 10,000 families. However, there is an absence of scientific evaluations of programme effectiveness. This study aims to fill this evidence gap, and the findings will be used to inform future modification, replication, and dissemination of the programme in other parts of China. This study will also contribute to the literature on the effectiveness of parent training programmes for ASD and for families living in low- and middle-income countries.

Methods A quasi-experimental design with a mixed-methods approach will be used, involving two consecutive waves of delivery of the SREIA programme. Parent participants will complete demographic and outcome questionnaires at baseline, immediate post-intervention, and 1- or 1.5-year post-intervention (conditional to funding). The implementation components will be assessed by collecting attendance and engagement registry data, facilitators filling out fidelity checklists, research staff observing programme sessions, and parents answering a satisfaction questionnaire. After the programme, some parents, facilitators, and NGO (non-governmental organisation) managers will be invited to take part in qualitative interviews or focus group discussions so as to explore their views about the programme, and to better understand the quantitative data obtained.

ELIGIBILITY:
The recruitment criteria for parents/primary caregivers from families with children with ASD will follow the existing strategies used by of the implementation organisation. Each primary caregiver will have one child participating in the program. Participating primary caregivers will be those who:

* Aged 18 or older,
* Undertake the responsibility for the daily care of a child between the ages of 3 and 6 years for at least 5 days a week,
* target child meets the diagnostic criteria for Autism Spectrum Disorder according to DSM-V (Diagnostic and Statistical Manual of Mental Disorders, 5th Edition); otherwise, an official letter of ASD diagnosis should be provided, and
* Provide informed consent to participate in the research.

Facilitator Inclusion Criteria:

* Aged 18 or older,
* Employees of the implementation organisation,
* Participate in the delivery of the program during this study, and
* Provide informed consent to participate in the research.

Program Manager Inclusion Criteria:

* Aged 18 or older,
* managers of the program, and
* Provide informed consent to participate in the research.

Parent/Primary Caregiver Exclusion Criteria:

* Parents/primary caregivers will be excluded if the child has been diagnosed with Cerebral Palsy. There will be no additional exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Change in frequency of child ehavioral problems | Differences between groups within 1 month after the end of intervention
  Child behavioral problems will be assessed using the Externalizing scale of the Child Behavior Checklist (CBCL) for Ages 1.5-5. The Externalizing scale measures child attention problems and aggressive behaviors using 24 items rated by parents based on child performance during the previous two months with a 3-point -type scale. The study will use the CBCL 1.5-5 for all families whose children will be between three to six years old. Lower scores suggest fewer behavioral problems. Research has shown sufficient test-retest reliability, internal consistency, convergent validity, and cross-cultural validity of CBCL 2-3 and CBCL 4-18 in China, but the evidence regarding the validity and reliability of this new version of CBCL 1.5-5 is currently limited. However, the CBCL 1.5-5 has shown good factorial validity among Chinese girls adopted into North American families; it has also demonstrated good internal validity with children with ASD.

SECONDARY OUTCOMES:
Change in frequency of ASD symptoms | Differences between groups within 1 month after the end of intervention
  ASD symptoms will be assessed using the Chinese version of the Autism Treatment Evaluation Checklist (ATEC), which comprise four subscales to measure child speech/language/communication, sociability, sensory/cognitive awareness, and health/physical/behavior. The scale has 77 items that are scored by parents. The health/physical/behavior subscale is rated using a 0 (not a problem)-to-3 (serious problem) point scale, whereas the other three subscales are rated using a 0 (not true)-to-2 (very true) point scale. Higher scores represent more ASD symptoms.
Change in frequency of parenting style: over-reactivity | Differences between groups within 1 month after the end of intervention
  Over-reactivity parenting style will be measured using the Over-Reactivity subscale (5 items) of the Arnold-O'Leary Parenting Scale (PS). The PS assesses dysfunctional discipline practices reported by parents using a 7-point Likert-type scale. Higher scores indicate more dysfunctional parenting practices.
Change in frequency of parenting style: supportive behaviors | Differences between groups within 1 month after the end of intervention
  Supportive parenting style will be measured using the Supporting Positive Behavior subscale (7 items) of the Parenting Young Children Scale (PARYC). The PARYC Supporting Positive Behavior subscale is rated by parents from 1 to 7 regarding the frequency with which they engaged in such parenting strategies during the last month. Higher scores represent more positive and proactive parenting practices. Higher scores indicate more supportive parenting practices.
Change in frequency of parental mental health symptoms | Differences between groups within 1 month after the end of intervention
  Parental mental health will be assessed using the Depression Anxiety Stress Scale-21 items (DASS-21), which consists of three self-report subscales (depression, anxiety, and stress) with each having 7 items that are rated from 0 (not apply to me) to 3 (apply to me very much or most of the time). Higher scores indicate a worse emotional state.
Change in family function | Differences between groups within 1 month after the end of intervention
  Family function will be assessed using the Chinese version of the Family APGAR scale, which consists of 5 items that are rated from 0 (never) to 2 (often) to examine the five functional components of adaptability, partnership, growth, affection, and resolve. Higher scores indicate that parents are more satisfied with their relationships with other family members.
Change in parental knowledge | Differences between groups within 1 month after the end of intervention
  Parental knowledge will be measured using of a questionnaire designed for the SREIA evaluation to assess parental understanding of ASD and child behaviors.

OTHER OUTCOMES:
Parent satisfaction: questionnaire | Within 1 month after the end of intervention
  Parent satisfaction will be assessed at post-intervention only using a questionnaire based on the Incredible Years® Autism Programme End-of-Course Satisfaction Questionnaire and tailored to the SREIA programme and Chinese context. The questionnaire covers a range of topics including overall impression; teaching format; information and techniques; facilitators; and parent groups. It consists of 30 items rated with a 3-point Likert-type scale. High scores represent higher levels of satisfaction.
Participant involvement | During the intervention
  The level of participant involvement will be captured by calculating rates of attendance, engagement, and dropout. The attendance rate will be assessed with an attendance sheet, which will be reported by facilitators and collected once a day; engagement rate will be based on the percentage of families who complete assigned homework and tasks during the practice sessions, using an attendance and engagement registry; dropout rate will be calculated based on families who miss at least 10 days and are not able to provide post-intervention data.
Implementation fidelity | During the intervention
  Implementation fidelity will be measured using facilitator checklists. Facilitators will report whether they deliver the core components prescribed in the manual. The fidelity score will comprise the ratio of delivered components to prescribed components. Dosage will be calculated using hours of delivery.
Quality of delivery: survey | During the intervention
  Quality of delivery will be assessed by research staff observing parent group sessions and filling out a quality of delivery survey. It consists of 28 items rated with a 4-point Likert-type scale and additional space to provide qualitative comments. High scores represent higher quality of delivery.
Acceptability/involvement/implementation (parents/primary caregivers): semi-structured interview | Six months after the completion of intervention
  Qualitative individual interviews will be conducted with around 15 parents, with the final number depending on when data saturation is reached. A semi-structured interview schedule will be developed to guide the interviews. The interview will cover the following topics: 1) understanding and use of skills, 2) perceived changes, 3) barriers to, facilitators of, and strategies to overcome the challenges of participation and engagement in the programme, and 4) acceptability and appropriateness of programme delivery and contents.
Acceptability/implementation (facilitators): semi-structured interview | Within 1 month after the end of intervention
  Focus groups will be conducted with around ten SREIA facilitators. A semi-structured interview schedule will be developed to guide the interviews. The discussion will cover the following topics: 1) barriers to, facilitators of, and strategies to overcome the challenges of program implementation, and 2) acceptability and appropriateness of program delivery and contents.
Acceptability/implementation/sustainability | Within 1 month after the end of intervention
  Qualitative individually interviews will be conducted with five program managers. he interviews with program managers will be structured to probe five dimensions that affect intervention impact including reach, effectiveness, adopt, implementation, and maintenance (RE-AIM).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Stars and Rain Education Institute for Autism, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data will not publicly available due to ethical requirements in the University of Oxford but will be available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Fang Z, Lachman JM, Qiao D, Barlow J. Controlled Trial of a Short-term Intensive Parent Training Program within the Context of Routine Services for Autistic Children in China. Psychosoc Interv. 2022 May 13;31(2):121-131. doi: 10.5093/pi2022a9. eCollection 2022 May. PMID 37360058